CLINICAL TRIAL: NCT03367351
Title: Web-Based Intervention Designed to Educate and Improve Adherence Through Learning to Use Continuous Glucose Monitoring
Acronym: IDEAL CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFT1DCGM2017; IRB201701822 (Other: University of Florida)
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Type 1 Diabetes Mellitus; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, un-blinded intervention/control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web-Based Educational Intervention (Experimental): Participants receiving the Web-Based Educational Intervention will be enrolled to the research protocol for six weeks of module-based learning and online discussion sessions and followed for a total of 3-months post CGM implementation to collect study measures.
  Interventions: Behavioral: Web-Based Education; Behavioral: Social Support
- Standard of Care (Placebo Comparator): Participants will receive standard clinical care. Similar study measures will be collected to compare between groups.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Web-Based Education — Completion of a CGM specific web-based educational intervention that includes a series of online learning modules.
  Arms: Web-Based Educational Intervention
Behavioral: Social Support — Engagement in peer-led CGM specific discussion boards
  Arms: Web-Based Educational Intervention
Behavioral: Standard of Care — Standard of Care - serves as the control group for the treatment arm
  Arms: Standard of Care

SUMMARY:
The goal of this pilot study is to produce a high-quality, theory-driven, therapeutic, web-based intervention that provides extended training and peer support to adolescents and young adults with type 1 diabetes who are newly implementing CGM. Overall, this web-based intervention represents an efficient way to bring together professionally-supported CGM educational materials and social support to overcome known barriers and address factors associated with inconsistent CGM use.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read and speak English
2. Diagnosed with type 1 diabetes (T1D) for > 3 months before consent is obtained
3. Aged >15 years and <24 years at time of enrollment
4. Must have access to a smartphone, tablet or laptop/desktop computer with high speed internet access and speaker
5. Must be using/initiating a Dexcom CGM

Exclusion Criteria:

1. Cognitive or learning disability (e.g., inability to read) that would preclude their ability to comply with the study protocol
2. Significant medical comorbidity in the adolescent or young adult that could, in the opinion of the PI, affect subject's capacity to follow study protocol
3. Previous use of a CGM within the last 3 months
4. Unwilling or unlikely to return to clinic for a follow-up HbA1c test
5. Unwillingness to accept randomization

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Adherence to CGM | 3 months
  Analyzing CGM data to determine if there is a difference in adherence between treatment and control group

SECONDARY OUTCOMES:
HbA1c | 1-week run in, 3-months post implementation
  The hemoglobin A1c value is a biologic measure of the glycemia that is the gold standard measure of "control" of diabetes. Collected through a blood sample.
CGM Satisfaction | 1-week run in, 7 weeks
  Survey instrument that measures self-reported satisfaction with CGM use
CGM Self-Efficacy | 1-week run in, 7 weeks
  Survey instrument that measures self-reported self-efficacy related to CGM use

CONTACTS AND LOCATIONS:
Overall Officials: Madison B Smith, BSN, PhD Candidate, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith MB, Albanese-O'Neill A, Yao Y, Wilkie DJ, Haller MJ, Keenan GM. Feasibility of the Web-Based Intervention Designed to Educate and Improve Adherence Through Learning to Use Continuous Glucose Monitor (IDEAL CGM) Training and Follow-Up Support Intervention: Randomized Controlled Pilot Study. JMIR Diabetes. 2021 Feb 9;6(1):e15410. doi: 10.2196/15410. PMID 33560234